CLINICAL TRIAL: NCT00311077
Title: Pharmacodynamic and Pharmacokinetic Properties of Insulin Glulisine (Apidra) in Comparison to Insulin Lispro (Humalog) in Healthy Lean and Obese Subjects
Brief Title: Insulin Glulisine in Healthy Lean and Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HMR1964A_1502
Record Dates: First submitted 2006-03-02; First posted 2006-04-05 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin glulisine

INTERVENTIONS:
Drug: Insulin Glulisine

SUMMARY:
Primary objective

* To investigate pharmacodynamic and pharmacokinetic parameters after s.c. administration of two different doses (low dose, 0.2 IU/kg and high dose, 0.4 IU/kg) of insulin glulisine across healthy subjects in 4 different BMI-classes (lean, overweight, moderately obese, severely obese), using the euglycemic clamp technique with the Biostator™.

Secondary objective

* To investigate the pharmacodynamic and pharmacokinetic properties after subcutaneous administration of insulin glulisine in comparison to insulin lispro and to investigate the safety and tolerability after subcutaneous administration of insulin glulisine in comparison to insulin lispro.

ELIGIBILITY:
Inclusion criteria :

* Normal HbA1c
* Women have to either be postmenopausal, surgically sterilized, or not pregnant and using adequate contraception.

Exclusion criteria :

* Systemic concomitant medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the serum insulin glulisine concentration and insulin lispro concentration | During the Study Conduct

SECONDARY OUTCOMES:
To measure blood glucose | During the study conduct
To measure glucose infusion rate | During the study conduct
To measure the serum C-peptide | During the study conduct
Adverse events collection | from the inform consent signed up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, MD, Study Director — Sanofi